CLINICAL TRIAL: NCT07023952
Title: Effect of Phenol Addition to Laser Treatment on Epithelialization and Healing Process in Pilonidal Sinus: A Prospective Randomized Controlled Clinical Trial
Brief Title: Effect of Phenol Addition to Laser Treatment on Epithelialization and Healing Process in Pilonidal Sinus
Acronym: PLEPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSL-FENOL-2025-001
Record Dates: First submitted 2025-06-08; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pilonidal Sinus Disease; Laser Therapy
Keywords: Minimally Invasive Treatment; Day Surgery
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: Two parallel groups: Group A receives laser treatment only, Group B receives combined phenol and laser treatment
Masking Description: Open-label study due to the nature of surgical interventions which cannot be blinded to participants or care providers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Treatment Only (Active Comparator): Participants receive laser treatment (SiLaC - Sinus Laser Closure) under local anesthesia. The pilonidal sinus area is cleaned, sinus openings are evaluated, and laser probe is inserted into sinus channels for ablation. Standard post-operative wound care is provided with same-day discharge.
  Interventions: Procedure: Laser Treatment
- Crystallized Phenol (Experimental): Participants receive combined treatment under local anesthesia. First, the pilonidal sinus area is cleaned and curetted, then crystallized phenol is applied into sinus channels. After a specified time, phenol is neutralized with normal saline, followed by laser treatment (SiLaC) application. Standard post-operative wound care is provided with same-day discharge.
  Interventions: Procedure: Laser Treatment; Drug: Crystallized Phenol

INTERVENTIONS:
Procedure: Laser Treatment — Minimally invasive laser ablation procedure performed under local anesthesia for pilonidal sinus treatment. Laser energy is delivered through a fiber optic probe inserted into the sinus tract to achieve thermal ablation of the sinus cavity.
  Other Names: Pilonidal Sinus Laser Ablation
Drug: Crystallized Phenol — rystallized phenol is applied directly into the pilonidal sinus channels after cleaning and curettage. The phenol remains in contact for a specified duration before being neutralized with normal saline irrigation.
  Other Names: Phenol Crystals
  Arms: Crystallized Phenol

SUMMARY:
This study compares two treatment approaches for pilonidal sinus disease: laser treatment alone versus laser treatment combined with phenol application. Pilonidal sinus is a common condition that affects young adults and can cause significant discomfort and time off work.

Participants will be randomly assigned to receive either laser treatment only (Group A) or laser treatment plus phenol application (Group B). Both treatments are minimally invasive and performed under local anesthesia as day surgery procedures.

The main goal is to determine if adding phenol to laser treatment speeds up the healing process (epithelialization) and improves patient outcomes. We will measure healing time, pain levels, return to daily activities, and quality of life over a 3-month follow-up period.

This research may help develop more effective treatment protocols that reduce healing time and improve patient comfort for people with pilonidal sinus disease.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical trial investigates whether adding crystallized phenol to laser treatment improves epithelialization and healing outcomes in patients with pilonidal sinus disease. The study will be conducted at Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital.

Study Design: 130 patients meeting inclusion criteria will be randomly assigned using computer randomization to two treatment groups (65 patients each):

Group A: Laser treatment only using SiLaC (Sinus Laser Closure) technique Group B: Combined phenol application followed by laser treatment

Treatment Procedures:

Group A receives local anesthesia, pilonidal sinus area cleaning, assessment of sinus openings, and laser probe application into sinus channels.

Group B receives local anesthesia, sinus area cleaning and curettage, crystallized phenol application into sinus channels, neutralization with saline after a specified time, followed by laser treatment.

Both groups receive standard post-operative wound care instructions and same-day discharge.

Follow-up Schedule:

Preoperative assessment Postoperative visits at 2 weeks, 4 weeks, and 3 months Clinical examination for epithelialization status Pain assessment using Visual Analog Scale (VAS 0-10) Quality of life evaluation using SF-36 questionnaire

Statistical Analysis: R software will be used for statistical analysis. Student's t-test or Mann-Whitney U test for continuous variables, chi-square test for categorical variables, and paired t-test for pre/post-treatment comparisons. Statistical significance set at p<0.05.

Primary Outcome: Time to complete epithelialization Secondary Outcomes: Postoperative pain scores, return to daily activities time, patient satisfaction, quality of life scores, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Primary pilonidal sinus disease
* Three or fewer pit counts
* Willing to participate in the study and signed informed consent form
* Able to attend follow-up visits

Exclusion Criteria:

* Age under 18 years
* More than three pit counts
* Acute abscess presentation
* Bilateral lateral extension
* Recurrent pilonidal sinus disease
* Immunocompromised patients
* Patients unable to attend follow-up visits
* Pregnancy (if applicable)
* Severe comorbidities that contraindicate surgery under local anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Time to Complete Epithelialization | From date of surgery until complete epithelialization is achieved, assessed up to 3 months
  Time required for complete epithelialization of the pilonidal sinus wound, assessed by clinical examination during follow-up visits. Complete epithelialization is defined as full closure of the wound with healthy epithelial tissue covering the entire treated area.

SECONDARY OUTCOMES:
Postoperative Pain Scores | Measured at 2 weeks, 4 weeks, and 3 months post-surgery
  Pain intensity measured using Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst pain imaginable)
Return to Daily Activities Time | From date of surgery until return to normal activities, assessed up to 3 months
  Time required for patients to return to normal daily activities and work, measured in days from surgery
Complication Rate | From surgery through 3 months follow-up
  Incidence of post-operative complications including infection, wound dehiscence, bleeding, or other adverse events
Patient Satisfaction- VAS score Patient Satisfaction Patient Satisfaction | At 3 months post-surgery
  Patient satisfaction measured using Visual Analog Scale (VAS) ranging from 0 (completely dissatisfied) to 10 (completely satisfied), where higher scores indicate better satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Sehit Prof. Dr. Ilhan Varank Training and Research Hospital, Istanbul, Other, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No